CLINICAL TRIAL: NCT01664884
Title: Internalized Stigma in a Sample of Young Adults With Bipolar Disorder or Schizophrenia.
Brief Title: Internalized Stigma in Patients With Bipolar Disorder or Schizophrenia
Acronym: ESTINT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Ricardo Alberto Moreno, University of Sao Paulo
Other Study IDs: ESTINT
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Stigma
Keywords: INTERNALIZED STIGMA; INSIGHT; SOCIAL ADEQUACY; BIPOLAR DISORDER; SCHIZOPHRENIA
MeSH Terms: conditions — Social Stigma; Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bipolar Disorder Patients: Bipolar Disorder Patients, with age between 18 to 40 years old, at euthymic phase.
- Schizophrenia Patients: Schizophrenia Patients, with age between 18 to 40 years old, with minimum or none positive symptoms.

SUMMARY:
The aim of this study is to explore the levels of internalized stigma in a sample of young patients with bipolar disorder or schizophrenia.

DETAILED DESCRIPTION:
The stigma is considered by patients, government organizations and health professionals a key point in mental illness (Griffiths et al, 2006). The related literature has focused on individuals with schizophrenia although there are indications that stigma act negatively in patients with bipolar disorder; this, in turn, is described in a few studies, always with heterogeneous samples, chronic and symptomatic patients (Perlick et al, 2001). It is also known that there is a significant association between affective symptoms and the presence of stigma, (Vázquez et al, 2010).

There are reports of higher levels of public stigma towards people with schizophrenia, compared to patients with bipolar disorder or unipolar depression, however there are no studies available on internalized stigma in such samples, especially in remitted patients . Since schizophrenia coexists with significant impairment of insight, such individuals may exhibit more difficulty internalizing the external bias and stereotypes. On the other hand, patients with bipolar disorder - despite being less discriminated by the public in relation to schizophrenia - probably have a high potential for self-stigma and its fearsome consequences, justified by higher levels of insight.

The investigators would like to examine whether the lower impairment of insight in young bipolar patients(in relation to young people with schizophrenia) could be accompanied by an increase in internalized stigma in this sample. It´s an observational, cross-sectional study with no intervention.

Hypothesis: the internalized stigma in young adults with bipolar disorder is identical to that of young patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder and schizophrenia according to DSM-IV-TR, presenting in euthymia (bipolar disorder) or without positive symptoms (schizophrenia), based on clinical assessment and confirmed by structured clinical interview SCID-P
* Age between 18 and 40 years
* Literate and able to understand the tasks required.
* Residents of Greater Sao Paulo.
* Patients and / or legal representatives must understand the nature of the study and sign an informed consent.

Exclusion Criteria:

* Patients with Schizoaffective Disorder or Mental Retardation.
* Unstable serious diseases including kidney disease, gastroenterology, respiratory, cardiovascular, endocrine, neurological, immunological or haematological.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The group will consist of patients from the Institute of Psychiatry, Hospital das Clinicas, Faculty of Medicine, University of São Paulo (HCFMUSP) diagnosed by DSM-IV-TR bipolar disorder (in remission) or schizophrenia (absence of positive symptoms).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alberto Moreno, MD PhD, Study Director — University of Sao Paulo
Locations (1):
- PROGRUDA-Institute of Psychiatry- HCFMUSP, São Paulo, São Paulo, Brazil